CLINICAL TRIAL: NCT07309965
Title: Feasibility Study on the Implementation of Local Muscle Vibration as Part of a Rehabilitation Program for Elderly Patients Following Fracture of the Upper End of the Femur
Brief Title: Feasibility of Integrating Local Vibration Into Rehabilitation of Elderly Patients After Hip Fracture
Acronym: ORTHOBOOSTER-P
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL24_1080
Record Dates: First submitted 2025-09-16; First posted 2025-12-30 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-12

CONDITIONS: Fracture Femur; Elderly
Keywords: Rehabilitation; Fracture of the upper end of the femur; Local muscle vibration; Geriatrics
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Intervention Model Description: A single-centre, prospective feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects aged 75 and over with surgery following a fracture of the upper end of the femur (Experimental): Patient, aged 75 and over, hospitalised in Medical and Rehabilitation Care no later than D14 of his operation for a fracture of the upper end of the femur
  Interventions: Diagnostic Test: Initial Assessment; Device: Standard rehabilitation programme combined with local vibration sessions; Other: Final assessment; Other: Acceptability and satisfaction questionnaire

INTERVENTIONS:
Diagnostic Test: Initial Assessment — Upon entering the SMR service, the patient receives several evaluations from the nurse.
  * a functional assessment :
    * Basic ADLs (BADLs) 6-point score
    * Instrumental ADLs (IADLs) 8-point score
  * a frailty assessment
  * a nutritional assessment
    * Body Mass Index (BMI)
    * Bioelectrical Impedance Analysis
    * JAMAR Grip Strength Test
  * A measurement of the maximum isometric strength of the non-injured limb (T0)
  * An assessment of physical performance using the Short Physical Performance Battery (SPPB)
  * An assessment of the risk of falling using TINETTI
  It has two subscales:
  * Balance section (maximum 16 points) Assesses sitting balance, sit-to-stand, standing balance, response to mild pushes, turning, etc.
  * Gait section (maximum 12 points) - Pain assessment using a simple verbal scale (EVS)
Device: Standard rehabilitation programme combined with local vibration sessions — The patient will receive a standard rehabilitation programme combined with local vibration sessions 5 times a week for 30 minutes each for 4 weeks.
  A record of these sessions will be completed every day by the rehabilitation specialist.
Other: Final assessment — The patient will undergo the same tests as the initial assessment, with the addition of a measurement of the isometric force on the injured limb (T1).
Other: Acceptability and satisfaction questionnaire — An acceptability and satisfaction questionnaire will be given to all the paramedical teams and patients who took part in the study in order to assess the potential constraints linked to the implementation.

SUMMARY:
Fractures of the upper end of the femur in elderly patients are the 2nd most common fracture.

A fracture leads to a syndrome of psychomotor maladjustment, encouraged by pain and aggravated by hospitalisation. In 2014, 50,000 women and 16,000 men suffered this type of fracture every year. The consequences are serious, with a one-year mortality rate of 20 to 24% and an institutionalisation rate of 25%. In 2015, the direct cost of hip fracture in France was estimated at around €1 billion.

In line with the recommendations of the National Institute for Health and Care Excellence (NICE) and the results of meta-analyses, it is recommended that, in the absence of surgical or medical contraindications, patients should be assessed within 24 hours of hip fracture surgery, with a view to initiating early mobilisation and multidisciplinary rehabilitation.

It has been shown in healthy subjects that prolonged application of localised vibrations optimises nerve capacity, leading to an increase in maximum voluntary force.

For population of frail elderly post-operative patients, this localised vibration technique could accelerate and improve functional recovery, particularly in terms of muscle strength, joint mobility and pain. A reduction in muscle loss is hoped for, with benefits in terms of tolerance compared with neurostimulation.

As part of the implementation of the above-mentioned recommendations, the investigators wish to assess the quality of the integration of this technique, already in use in the department on an ad hoc basis, into the organisation of the department and of the patient's care pathway as a complement to the rehabilitation protocols, by identifying the obstacles and facilitating factors. The study will also provide the first estimates of the effect on muscle recovery.

The investigator hypothesise that this local vibration protocol can be integrated into the rehabilitation department's work schedule and into the patient's care pathway, and that it will be acceptable to both the patient and the nursing staff.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 75 or over who have undergone surgery for a fracture of the upper end of the femur
* Hospitalised in the SMR department no later than D14 of their operation
* Resource Iso Group greater than or equal to 3 on the Aggir scale
* Patient capable of consenting who has signed a consent form or patient unable to express consent at the discretion of the principal investigator, informed and not opposed to the study, for whom a trusted person, or if not available, the family, or if not available, a close relative has signed an informed consent within a maximum of 2 days. For patients under guardianship, the guardian's consent will be requested, and for patients under curatorship, the patient will sign the consent in the presence of the curator within a maximum of 2 days as well.
* Affiliated to a social security scheme

Exclusion Criteria:

* Persons deprived of their liberty by a judicial or administrative decision
* Individuals with severe psycho-behavioral disorders (major psychiatric or neurocognitive disorders)
* Persons admitted to a health or social establishment for purposes other than research
* Contraindications to electrical stimulation:

  * Patient with active devices such as pacemakers, defibrillators, insulin pumps, neurostimulators, etc
  * Patient with phlebitis or risk of thrombosis
  * Epileptic patient
  * Patient with fragile skin or open wounds on the lower limbs
* Subject participating in another interventional study with an exclusion period still in progress at pre-inclusion.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2026-11-19 (Estimated); Study Completion 2026-12-19 (Estimated)

PRIMARY OUTCOMES:
Feasibility of implementing local muscle vibration sessions | Week 4 : End of standard rehabilitation protocol plus local vibrations
  Completion of local muscle vibration sessions. The operation will be considered complete if 5 sessions lasting 30 minutes per week have been carried out for 4 weeks.

SECONDARY OUTCOMES:
Number of eligible patients not taking part in the study | Week 4 : End of standard rehabilitation protocol plus local vibrations
  Number of eligible patients not participating in the study and description of reasons
Reasons for not completing sessions and incomplete completion of sessions | Week 4 : End of standard rehabilitation protocol plus local vibrations
  Description of the reasons why sessions were not carried out (less than 5 sessions) and why sessions were not carried out in full (less than 30 min) over 4 weeks of rehabilitation using a local vibration session traceability sheet.
Tolerability of the muscle vibration technique in real-life care conditions | Week 4 : End of standard rehabilitation protocol plus local vibrations
  Description of the effects noted during the local vibration sessions (redness, heat, pain or other discomfort) using the local vibration session traceability form.
Results after the local muscle vibration technique in terms of variation between the start of rehabilitation and after 4 weeks in following parameters: • Isometric strength (in %) | Week 4 : End of standard rehabilitation protocol plus local vibrations
  Isometric force differential (measured by the physiotherapist using a dynamometer).This differential (in %) is defined by the following equation:
  (FIM injured limb (T1) - FIM non-injured limb (T0)) / FIM non-injured limb (T0)
Results after the local muscle vibration technique in terms of variation between the start of rehabilitation and after 4 weeks of the rehabilitation programme in the following parameters: • Physical performance | At 4 weeks - End of standard rehabilitation protocol plus local vibrations
  • Clinically significant improvement in physical performance between the start of rehabilitation and after 4 weeks of the rehabilitation programme.
  Physical performance was assessed by the overall score of the SPPB (Short Physical Performance Battery), based on three components: walking speed, chair raising and balance tests. A global score of 0 to 6 is a low performance score, a global score of 7 to 9 is an intermediate performance score and a global score of 10 to 12 is a high performance score. An improvement will be considered clinically significant for patients who change performance group positively.
Evaluate the results after the local muscle vibration technique in terms of variation between the start of rehabilitation and after 4 weeks of the rehabilitation programme in the following parameters: • Risk of falling | At 4 weeks - End of standard rehabilitation protocol plus local vibrations
  A clinically significant reduction in the risk of falling between the start of rehabilitation and after 4 weeks of the rehabilitation programme.
  This risk of falling is assessed by the TINETTI score. A score of less than 20 points is a very high fall risk score, a score of 20 to 23 points is a high fall risk score and a score of 24 to 28 points is a low fall risk score. An improvement will be considered clinically significant for patients who change fall risk group positively.
Results after the local muscle vibration technique in terms of variation between the start of rehabilitation and after 4 weeks of the rehabilitation programme in the following parameters: • Transfers | At 4 weeks - End of standard rehabilitation protocol plus local vibrations
  Difference between the score obtained for transfers between the start of rehabilitation and after 4 weeks of the rehabilitation programme.
  Each type of transfer (lying>seated, sitting>standing, bed>chair) will be scored as follows 0: no assistance, 0.5: partial material and/or human assistance, 1: total assistance, 2: not feasible. These sub-scores will be added together to obtain an overall transfer score.
Evaluate the results after the local muscle vibration technique in terms of variation between the start of rehabilitation and after 4 weeks of the rehabilitation programme in the following parameters: • Pain | At 4 weeks - End of standard rehabilitation protocol plus local vibrations
  Difference in pain score between the start of rehabilitation and 4 weeks after the rehabilitation programme.
  Pain was assessed using a simple verbal scale (0: Absent, 1: Mild, 2: Moderate, 3: Intense, 4: Unbearable).
Measure patients' perceptions of the use of local muscle vibration in their rehabilitation protocol | At 8 weeks - End of protocol
  Evaluation scale (5-point Likert scale) measuring the patient's perception of the use of local vibration in their rehabilitation programme (comfort and ease of use, perceived effectiveness, and overall satisfaction). Collection of points for improvement. The higher the score, the more the patient agrees.
Measure the perception of healthcare professionals in the field regarding the use of local muscle vibration as part of their current functional rehabilitation protocol. | At 8 weeks - End of protocol
  Evaluation scale (5-point Likert scale) measuring nursing staff's perception of the use of local vibration in a rehabilitation programme (experience of use, ease of integration into practice, safety and tolerance, overall satisfaction). Collection of points for improvement. The higher the score, the more the patient agrees.

CONTACTS AND LOCATIONS:
Locations (1):
- HOPITAL PIERRE GARRAUD - Service de MEDECINE GERIATRIQUE, Lyon, France